CLINICAL TRIAL: NCT02714777
Title: General Anesthesia and Autonomic Nervous System in Children
Acronym: ANESPEDIA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608014; 2016-A00295-46 (Other: ANSM)
Record Dates: First submitted 2016-03-11; First posted 2016-03-21 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2016-05

CONDITIONS: Anesthesia, General
Keywords: General anesthesia; Autonomic nervous system; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric population from 4 to 8 years-old: Description of the Autonomic nervous system activity (parasympathetic activity)
  Interventions: Device: Autonomic nervous system activity

INTERVENTIONS:
Device: Autonomic nervous system activity — Autonomic nervous system activity (parasympathetic activity) will be measured by electrocardiogram (holter) during 24 hours postoperative

SUMMARY:
The objective of the ANESPEDIA study is to describe in a pediatric population (aged from 4 to 8 years old) receiving elective surgery, the impact of general anesthesia on autonomic nervous system and their kinetics of early postoperative course (24 hours).

DETAILED DESCRIPTION:
Some physiological factors such as sport activity or pathological as sepsis, certain chronic diseases or diabetes are known to modulate the overall autonomic activity and the intrinsic capacity of the individual to regulate its sympathovagal balance. These influences can alter the physiological autonomic balance sometimes with positive consequences on the Cardiac frequency-breathing control, blood pressure adjustment depending on the position of the individual, on the status of blood volume, but sometimes deleterious with bad regulation of sinus cardiac activity and respiration rate.

General anesthesia is recognized as one of the factors that can modify more or less sustainable the sympathovagal autonomic balance. While many studies described the effects of anesthesia on the autonomic nervous system, most data are done in adult subjects. For the child who sees intrinsically autonomic physiological changes related to its maturative status, assessment of the impact of anesthesia in the pediatric population in per and postoperative was never realized.

ELIGIBILITY:
Inclusion Criteria:

* Post-anesthesia Monitoring in pediatric intensive care units or Pediatric Surgery Hospital North of Saint Etienne.
* Compendium of the form signed by the holder of parental authority

Exclusion Criteria:

* Child with pathologies reaching the central nervous system or the brain stem.
* Children with a severe pathology of cardio-respiratory or heart being referred to treatment.
* Children requiring emergency surgery or trauma or septic or inflammatory context

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 4 to 8 years enjoying a scheduled surgery without any infection or trauma context and performed under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Description of parasympathetic activity evolution by heart rate variability | 24 hours
  Parasympathetic activity evolution will be described by heart rate variability

SECONDARY OUTCOMES:
Heart rate variability (HRV) | 24 hours
  HRV is measured by a 24H-Holter Electrocardiography (ECG). It is a composite outcome : SDNN, pNN30, pNN50, RMSSD, SD1, SD2, LF, VLF, LF/HF ratio and Ptot indexes
Heart rate variability (HRV) | at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24 Hours
  HRV is measured by a 24H-Holter Electrocardiography (ECG). It is a composite outcome : HF, SDNN, pNN30, pNN50, RMSSD, SD1, SD2, LF, VLF, LF/HF ratio and Ptot indexes

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No